CLINICAL TRIAL: NCT03629730
Title: Testing the Dose-response of Coordination Training for Older Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Kathleen Bell, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU 082017-078
Record Dates: First submitted 2018-08-08; First posted 2018-08-14 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Mobility Limitation
Keywords: coordination
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Intervention Model Description: Three intervention dose groups and one active control group will be compared.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The Principal Investigator and Research Coordinators conducting participant assessments will be masked as to participant group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High dose (Experimental): Will receive the greatest duration of coordination intervention training.
  Interventions: Behavioral: Coordination training
- Intermediate dose (Experimental): Will receive a moderate duration of coordination intervention training.
  Interventions: Behavioral: Coordination training
- Low dose (Experimental): Will receive a short duration of coordination intervention training.
  Interventions: Behavioral: Coordination training
- Active control (Active Comparator): Will perform the same number and duration of physical exercises as the High Dose group, but while moving one body segment at a time.
  Interventions: Behavioral: Coordination training

INTERVENTIONS:
Behavioral: Coordination training — The intervention will consist of 8 weeks of exercises to decrease the variability of participants' body and gait coordination. The intervention will consist of 1 training session /week in the Mobility Research Laboratory and 4 days of home-based training. In each session participants will perform 6 trials of 4 body coordination exercises and 1 gait exercise. In the intervention sessions participants will perform interlimb coordination exercises, synchronizing body segments with auditory metronome tones. Participants also will perform a gait exercise by synchronizing steps with an auditory metronome during walking. The metronome will assist participants to retrain their movement timing to decrease coordination variability.

SUMMARY:
There is an urgent need for interventions to reduce mobility limitations that affect over 15 million older adults and contribute to falls, disability, hospitalization and death. This training will give Dr. James the skills to become an independent researcher developing interventions to decrease mobility limitations, disability and falls in older adults. His multidisciplinary mentorship team, led by Kathleen Bell, MD, has extensive experience with externally sponsored research, expertise in the targeted training domains, mentoring new investigators, and is highly committed to Dr. James' development as a researcher.

Dr. James has identified novel impairments in rhythmic interlimb and gait coordination as strongly linked to mobility among community-dwelling older adults. Currently, no treatment for limb coordination exists. In an effort to advance the development of treatments for mobility limitations, the objective of the proposed research is to examine the dose-response of an innovative intervention to improve coordination in community-dwelling older adults with mobility limitations. The intervention uses a metronome to retrain coordination impairments that develop with age, and consists of practice improving the coordination of the right and left: a) ankles; b) shoulders; and c) ankles and shoulders, while lying supine, and d) the arms and legs during walking; by synchronizing movements with a metronome.

This project is significant in that the approach may offer a cost-effective, clinically applicable, and efficacious means of reducing mobility limitations in older adults. We will initially refine the intervention, and subsequently conduct a randomized trial of 2-, 4- and 8-week intervention treatments vs. physical activity control with (N=120) community-dwelling older adults aged >70 years with mobility limitations. These treatment durations correspond to what rehabilitative care providers would consider a short vs. medium vs. long duration (dose) of treatment. We will examine the magnitude and duration of change in interlimb ankle coordination and gait coordination for each group. We will estimate the coordination effect sizes for a minimal clinically important difference in mobility performance, and explore changes in upper limb coordination and performance-based and self-reported mobility.

DETAILED DESCRIPTION:
Concise Summary of Project:

The objective of the proposed research is to examine the dose-response of an intervention to improve interlimb and gait coordination in community-dwelling older adults with mobility limitations. The investigators will compare the effects of 3 doses of the intervention and a physical activity control. The intervention will consist of exercises for performing movement coordination patterns: 1) plantar flexing and dorsiflexing the right and left ankles; 2) flexing and extending the right and left shoulders; and 3) synchronizing the steps during walking with auditory metronome tones. Treatment will mirror outpatient rehabilitative care in that it will involve 1 weekly visit to the clinical laboratory and 4 days of home exercises each week, focusing on limb movement coordination. A physical activity control group will perform a similar treatment program of range of motion exercises that do not target coordination.

The treatment arms will consist of three doses of an intervention to improve coordination and a physical activity control arm. The three doses will consist of different durations of daily training in coordination exercises. Primary outcome variables are the standard deviation of relative phase of the ankles during rhythmic ankle coordination, and the Phase Coordination Index (a measure of gait coordination) during normal pace walking. Secondary outcomes will be the standard deviation of relative phase during rhythmic shoulder coordination, and Short Physical Performance Battery score. Key study endpoints will be at the end of the 8 week intervention, and 2-week follow up assessments up to 8-weeks post-intervention.

The maximum number of subjects to be consented, including projected screen failures and early withdrawals is 250. The study will last five years. Conditions that would result in subjects exiting the study prior to expected completion are death, moving away from the area, injury, the development of exclusionary comorbidities, safety reasons, and withdrawal of consent.

Study Procedures:

Recruitment Participants will be recruited through a letter mailed to addresses of individuals listed on the Dallas, Fort Worth, Irving, and Arlington, TX voter registration lists as being ≥ 70 years of age. Individuals potentially interested in participating in the study can contact the Principal Investigator (PI) or Research Coordinator (RC) at the telephone number or email provided in the letter.

Those who qualify for the study will be given a series of physical movement assessments and questionnaires. Participants will attend the research study once weekly for 10 weeks (2 weekly screening/baseline assessments, 8 weekly intervention sessions), followed by once every 2 weeks for another 8 weeks, for a total of 14 laboratory visits. The duration of each visit will be approximately 60 minutes. On the initial day of intervention or control training, participants will be scheduled for their subsequent days of weekly participation. In the event of an emergency the PI or RC will contact ext. 88911 (UTSW Emergency Services). In the event of a fall or other emergency and an ambulance must be called, while waiting for the ambulance to arrive our research personnel will provide assistance to the participant as instructed by the emergency operator. Participants will arrange for their own transportation to and from the laboratory.

Physical movement assessments The investigators will assess ankle and shoulder coordination by having participants lie down in a supine position on a physical therapy table and: a) plantar- and dorsi-flex their right and left ankles; and b) flex and extend their right and left arms (directly in front of them). The participants will perform 2 trials of 45 seconds duration of each task while synchronizing their movements with an auditory metronome we will play for them. A motion capture system will be used to collect 3-dimensional data on the body movement while participants perform the physical movement testing. This system is a set of infrared cameras on tripods that will be situated around participants. The camera system tracks the 3-D position of small reflective balls will be taped to the back of participants' arms, feet, head, and upper back. These reflective balls will be taped to elastic bands that will be wrapped around the participants' body. This camera system records infrared light and does not capture video images.

Participants will also walk 6-9 times across a 20 foot long walkway, with short rest breaks given between each pass across the walkway. The researcher will walk alongside (but off the walkway) the participant. The walkway is an instrumented mat that collects data from footfalls. This data will be used to assess gait patterns.

Participants will also perform the SPPB every 2 weeks when they come to the lab, using the same procedures as for exclusionary testing.

Questionnaires The participants will be asked a series of questions on their handedness and footedness (right or left), their race/ethnicity, years of education, annual family income, overall health, any chronic medical conditions, history of falling in the past 12 months, fear of falling, pain, and two connect-the-dot tests (Trail Making Tests A and B) that assess executive function. There are also a series of questions asked regarding participants' ability and frequency of performing physical activities (Late Life Function and Disability Instrument). These questionnaires are included in the IRB application materials.

The questionnaires will be administered during one of the first two days of screening/baseline assessments, at the end of the intervention (week 12), and on the last follow up session (week 22). The time for administration of the questionnaires will be approximately 40 minutes each day.

The total time for administering the physical testing will be approximately 20 minutes. The physical testing will be conducted on the first two screening/baseline testing sessions, every two weeks during the intervention (8 weeks), and every two weeks during the 8-week follow up testing. After completing the 2 screening/baseline testing sessions, participants will be randomly assigned to one of 4 groups: low, moderate, or high dose intervention; or physical activity control.

Participants will perform the intervention or physical activity control exercises in the Mobility Research Laboratory at UT Southwestern once per week for 8 weeks. During each training session the participants will practice rhythmically moving two parts of their body at a time. Each practice session will be approximately 30 minutes in duration, including rest breaks as needed by each individual. The participants will be instructed to make comfortable movements, to rest as needed and to stop moving if any movement causes them pain. Participants will be instructed on exercises they are to perform at home on 4 days of the subsequent week.

Intervention groups The rhythmic coordination exercises will be to synchronize the following body segments with auditory metronome tones. Exercises 1-4 will be performed supine; exercise 5 will be performed during walking

Body segments: Osteokinematic movement:

1. Right and left ankles Dorsiflexion-plantarflexion
2. Right and left shoulders (glenohumeral joints) Flexion-extension
3. Right shoulder (glenohumeral joint) and ankle. Flexion-extension with dorsiflexion-plantarflexion, respectively.
4. Left shoulder (glenohumeral joint) and ankle. Flexion-extension with dorsiflexion-plantarflexion, respectively.
5. Arms and legs during walking. Normal walking arm and leg swing.

Participants assigned to the low, moderate, and high dose intervention groups will practice synchronizing movements of their right and left ankles, right and left shoulders, and right and left steps with an auditory metronome. The researchers will provide participants with a take-home metronome for use during the exercises. These exercises will be varied slightly each week. This will be a very low impact type of training (it is designed to improve coordination, not endurance or strength).

The intervention will consist of 8 weeks of exercises to decrease the variability of participants' body and gait coordination. The intervention will consist of 1 training session /week in the Mobility Research Laboratory and 4 days of home-based training. In each session participants will perform 6 trials (of 30 seconds duration) of 4 body coordination exercises and 1 gait exercise (total duration approximately 30 minutes/session). In the intervention sessions participants will perform interlimb coordination exercises, synchronizing body segments with auditory metronome tones. Participants also will perform a gait exercise by synchronizing steps with an auditory metronome during walking around in their home. The metronome tone frequency will correspond with a percentage of the participant's normal walking cadence. The metronome will assist participants to retrain their movement timing to decrease coordination variability.

ELIGIBILITY:
Inclusion Criteria:

* Aged 70 years or older
* Walk 20 feet without personal assistance
* Sufficient vision to read written materials
* Sufficient hearing to synchronize movements with auditory metronome tones.

Exclusion Criteria:

* Severe language, visual, or hearing deficits
* Inability to perform the intervention exercises
* Self-report of:

A diagnosis or prescription of medications consistent with any psychiatric disorder Parkinson's disease Alzheimer's disease Stroke Severe head injury in the last two years A history of cardiovascular disease Having a terminal disease Major surgery or myocardial infarction in the past 6 months Planned major surgery Major medical problems interfering with safe and successful balance and walking Inability to read, speak and understand English Plan to leave the area within the next 1 year. Chronic pain that interferes with walking or standing

* The Short Physical Performance Battery score will be administered during the two baseline testing sessions. A score outside the range of 4-9 on either day will result in exclusion.
* 5.07/10-g monofilament testing will be conducted on the two baseline testing sessions to screen for clinically relevant neuropathy. A negative outcome on this test on either day will result in exclusion.
* Mini-Mental State Examination score <18

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 108 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Ankle coordination variability | Every 2 weeks from baseline until 8 weeks post-intervention.
  Change in the standard deviation of the relative phase between the ankles during rhythmic antiphase coordination synchronizing with a metronome.
Gait coordination | Every 2 weeks from baseline until 8 weeks post-interention.
  Change in the Phase Coordination Index of the right-left stepping pattern during normal pace walking.

SECONDARY OUTCOMES:
Short Physical Performance Battery | Every 2 weeks from baseline until 8 weeks post-intervention.
  Change in the composite score based on timed performances of normal walking speed, 5 repetition chair rise, and balance.
Shoulder coordination variability | Every 2 weeks from baseline until 8 weeks post-intervention.
  Change in the standard deviation of the relative phase between arms during rhythmic antiphase coordination while synchronizing with a metronome.

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No